CLINICAL TRIAL: NCT02186470
Title: Feasibility of Assessing Radiation Response With MRI/CT Directed Preoperative Accelerated Partial Breast Irradiation in the Prone Position for Hormone Responsive Early Stage Breast Cancer
Brief Title: Intensity Modulated Accelerated Partial Breast Irradiation Before Surgery in Treating Older Patients With Hormone Responsive Stage 0-I Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sasha Beyer, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-13282; NCI-2014-01248 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Estrogen Receptor-positive Breast Cancer; Invasive Ductal Breast Carcinoma; Invasive Ductal Breast Carcinoma With Predominant Intraductal Component; Medullary Ductal Breast Carcinoma With Lymphocytic Infiltrate; Mucinous Ductal Breast Carcinoma; Papillary Ductal Breast Carcinoma; Progesterone Receptor-positive Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Tubular Ductal Breast Carcinoma
Keywords: Breast Cancer; Early Stage Breast Cancer; Hormone responsive breast cancer
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Breast Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (image-guided intensity-modulated APBI) (Experimental): Patients undergo image-guided intensity-modulated APBI twice daily (BID) in the prone position over a period of 5-10 days for a total of 10 treatment. Within 4-6 weeks post-APBI, patients undergo lumpectomy.
  Interventions: Radiation: accelerated partial breast irradiation; Radiation: intensity-modulated radiation therapy; Radiation: image-guided radiation therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Radiation: accelerated partial breast irradiation — Undergo image-guided intensity-modulated APBI
  Other Names: APBI
Radiation: intensity-modulated radiation therapy — Undergo image-guided intensity-modulated APBI
  Other Names: IMRT
Radiation: image-guided radiation therapy — Undergo image-guided intensity-modulated APBI
Procedure: therapeutic conventional surgery — Lumpectomy

SUMMARY:
This pilot clinical trial studies intensity-modulated accelerated partial breast irradiation (APBI) before surgery in treating older patients with estrogen receptor positive or progesterone receptor positive stage I breast cancer. APBI is a specialized type of radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Giving radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Establish the feasibility for preoperative APBI delivered with IMRT in the prone position using daily CT guidance for Stage I breast cancer patients who are intended to undergo a lumpectomy for breast conserving therapy.

SECONDARY OBJECTIVES:

1. To determine the acute and late surgical and radiation toxicity of preoperative APBI delivered with IMRT in the prone position.
2. To document the cosmetic appearance of the breast when treated with preoperative APBI IMRT in the prone position.
3. Establish the percentage of patients that can meet dosimetric goals and normal tissue constraints if treated with preoperative APBI IMRT in the prone position.
4. Evaluate molecular changes in breast cancer and/or stroma before and after preoperative APBI

OUTLINE:

Patients undergo image-guided intensity-modulated APBI twice daily (BID) in the prone position over a period of 5-10 days for a total of 10 treatment. Within 4-6 weeks post-APBI, patients undergo lumpectomy.

After completion of treatment, patients are followed up at 4 weeks and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient must consent to be in the study and must have signed an approved consent form conforming with federal and institutional guidelines.
* Patient must be ≥ 50 years
* Core biopsy demonstrating breast cancer and receptors that are ER or PR positive.
* Core tissue must have HER 2 negative followed by current ASCO/CAP guidelines.
* The patient must have clinical node negative, stage I breast cancer.
* The surgical treatment must be intended to be a lumpectomy
* The biopsy site must have been demarcated by a clip(s)
* Gross disease must be unifocal on Mammo/ MRI imaging
* Patients must have estrogen receptor (ER) and progesterone receptor (PR) analysis performed on core biopsy
* Patient must be able to tolerate lying in the prone position with arms extended forward.
* Must be able to tolerate MRI scan with contrast
* At the time of enrollment, patients must have had bilateral mammograms within 6 months.
* Patients must be willing to undergo breast cancer surgery minimally 4, maximally 6 weeks post APBI.
* Patients with a history of non-breast malignancies are eligible if they have been disease free for 5 or more years prior to enrollment and are deemed by their physicians to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.

Exclusion Criteria:

* Age < 50 years
* Hormone unresponsive breast cancer
* T-2 ( > 3.0 cm), T-3, Stage III, or Stage IV breast cancer.
* N-1, N-2, or N-3 clinical axillary nodes
* Mastectomy intended
* Unwilling to undergo anti-endocrine therapy
* Suspicious microcalcification, densities, or palpable abnormalities ( in the ipsilateral or contralateral breast) unless biopsied and found to be benign.
* Non-epithelial breast malignancies such as sarcoma or lymphoma.
* Paget's disease of the nipple
* Proven multicentric carcinoma (invasive or DCIS) in more than one quadrant or separated by > 4 centimeters.
* Any prior treatment with radiation therapy, chemotherapy, biotherapy, or hormone therapy for the currently diagnosed breast cancer prior to study enrollment.
* Prior breast or thoracic RT for any condition.
* Psychiatric of addictive disorders or other condition that in the opinion of the investigator would preclude the patient from meeting the study requirements.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the reproducibility of the MRI directed preoperative APBI treatment method | 4-6 weeks post-APBI
  Acceptability of the definition of treatment targets by MRI, radiation virtual IMRT plans and completion of treatment (APBI and surgery).

SECONDARY OUTCOMES:
Acute surgical and radiotherapy toxicity as scored by the National Cancer Institute Common Toxicity Criteria (NCI CTCAE) version 4.0 | Up to 4 weeks post-surgery
Late surgical and radiotherapy toxicity as scored by the NCI CTCAE version 4.0 | Up to 5 years
Cosmetic outcome by the physician and patient | At year 1
Cosmetic outcome by the physician and patient | At year 3
In-breast recurrence | Up to 5 years
Regional recurrence | Up to 5 years
Distant metastases | Up to 5 years
Disease free survival | Up to 5 years
Overall survival | Up to 5 years
Exploratory evaluation of patient breast cancer tissue and serum for CSCs, biomarkers and miRNAs | Up to 4 weeks post-surgery
  Correlative analyses

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Beyer, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (2):
  • Informed Consent Form: Cohort 1 Informed Consent (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT02186470/ICF_000.pdf
  • Informed Consent Form: Cohort 2 Informed Consent (2025-07-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT02186470/ICF_001.pdf